CLINICAL TRIAL: NCT01786486
Title: AMPLATZER Cardiac Plug (ACP) Registry-Long Term Follow-up Protocol
Acronym: ACPR
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CL03562
Record Dates: First submitted 2013-01-29; First posted 2013-02-08 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Delivery system entry
  Interventions: Device: Amplatzer Cardiac Plug

INTERVENTIONS:
Device: Amplatzer Cardiac Plug

SUMMARY:
The objective of the AMPLATZER Cardiac Plug (ACP) Registry Long Term Follow-up study is to evaluate long term performance of the ACP in closure of the Left Atrial Appendage (LAA) in subjects with nonvalvular atrial fibrillation and assess adverse events up to two (2) or more years post implant.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a documented history of paroxysmal, persistent or permanent nonvalvular atrial fibrillation (documentation may include an electrocardiogram (ECG), Holter, or event recorder)
* Subject must be ≥18 years of age

Exclusion Criteria:

* Subject with an implanted atrial septal defect (ASD) device or patent foramen ovale (PFO) device
* Subject who has a history of surgical ASD or PFO repair
* Subject with a history of stroke and unrepaired PFO
* Subject who has moderate to severe aortic or mitral valve stenosis or regurgitation as assessed by the investigator
* Subject who has a mitral or aortic prosthetic valve
* Subject who has a planned ablation procedure for atrial fibrillation 30 days after the ACP implant
* Subject with New York Heart Association (NYHA) grade 4
* Subject with evidence of pericardial effusion at baseline evaluation
* Subject who has complex atheroma with mobile plaque of the descending aorta and/or aortic arch
* Subject who has an intracardiac thrombus
* Subject who has carotid disease as assessed by the investigator, requiring treatment, which includes revascularization and/or medical treatment
* Subject with active infection or active endocarditis
* Subject who has an acute or recent myocardial infarction (MI) or unstable angina (recent is defined as within 6 months of implant date)
* Subject who has had recent major cardiac surgical procedure (recent is defined as within 6 months of implant date)
* Subject with malignancy or other illness where life expectancy is less than one year
* Subject who is pregnant, breastfeeding, or desires to become pregnant during their first six months of follow-up
* Subject or legally authorized representative who is unable to provide informed consent
* Subject who will not be able to be followed for the duration of the clinical study
* Subject with any medical disorder or severe disability that would interfere with completion or evaluation of clinical study results (for e.g. uncontrolled hypertension, uncontrolled diabetes, renal failure, in situ inferior vena cava (IVC) filter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2009-08; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The rate of occurrence for any reported adverse event experienced by subjects enrolled. | Through 2 years
Closure | 6 months
  Defined as absence of flow or flow of ≤3mm jet into the LAA at procedure and at six (6) months as assessed by Transoesophageal Echocardiography (TOE).
Technical success | At implant
  Defined as delivery and release of the ACP device, including recapture and/or replacement, as necessary. This success will be calculated among subjects in whom the device enters the body

CONTACTS AND LOCATIONS:
Locations (15):
- Hospital Na Homolce Cardiocentrum, Prague, Czechia
- Germany (7):
  - St. Marien-Hospital Bonn, Bonn
  - University of Bonn, Bonn
  - Cardiovascular Center Frankfurt, Frankfurt
  - Kardiocentrum Frankfurt an der Klinik Rotes Kreuz, Frankfurt
  - University Medicine Goettingen, Göttingen
  - Asklepios Kliniken GmbH/Asklepios Klinik Harburg, Hamburg
  - Stadt Krankenhaus Pirmasens gGmbh, Pirmasens
- Mater Misericordiae University Hospital, Dublin, Ireland
- Spain (4):
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 'Virgen de la Arrixaca", Murcia
  - Hospital de Navarra, Pamplona
- United Kingdom (2):
  - Royal Sussex County Hospital-UK, Brighton
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Manuscript has been submitted to Euro Intervention Sept 2016